CLINICAL TRIAL: NCT04170231
Title: Bleeding in Critically Ill Children With Underlying Oncologic Diagnoses
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-407
Record Dates: First submitted 2019-11-19; First posted 2019-11-20 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Bleeding
Keywords: Critically Ill Children; 19-407
MeSH Terms: conditions — Neoplasms; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"Bleeding in Critically Ill Children with Underlying Oncologic Diagnoses ," will be a prospective observational cohort study looking at the epidemiology of bleeding in the pediatric ICU population at MSK.

ELIGIBILITY:
Inclusion Criteria:

* All children (≥28 days old through 18 years of age) with an oncologic diagnosis admitted to the PICU at Memorial Sloan Kettering Cancer Center
* An oncologic diagnosis will include those with a cancer diagnosis or those being treated at MSK for blood disorders, immunodeficiencies and complications of transplant.

Exclusion Criteria:

* Preterm infants (<44 weeks gestation at age of enrollment) as in these patients most bleeding etiologies are specific to the neonatal period and the bleeding assessment tool is not calibrated for this population
* Known limitation of care at enrollment (standing Do Not Resuscitate order), as the interventions and clinical outcome would be biased
* Pre-existing bleeding disorders

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All subjects admitted to the pediatric ICU at MSKCC will be included in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
the incidence of severity of bleeding | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Nellis, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm